CLINICAL TRIAL: NCT06069037
Title: Sequential Adult Left Lateral Lobe Liver Transplantation for Patients With Early Acute on Chronic Liver Failure: a Single Center, Prospective, Single Arm Study
Brief Title: SALT for Treatment of Patients With Early ACLF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-183-C
Record Dates: First submitted 2023-09-25; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Sequential Adult Liver transplantation; Left lateral segment; Portal inflow modulation; Acute-on-chronic liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: SALT for patients who meet the enrollment conditions and successfully match the donor liver. Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SALT surgery (Experimental): SALT for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume
  Interventions: Procedure: sequential adult left lateral lobe liver transplantation (SALT)

INTERVENTIONS:
Procedure: sequential adult left lateral lobe liver transplantation (SALT) — SALT for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.

SUMMARY:
ACLF is a syndrome characterized by rapid deterioration of liver function in chronic liver disease or undiagnosed chronic liver disease, with a high risk of short-term death. Both CMA and EASL mentioned that there is currently lack of specific drugs and treatment of liver failure. For patients with ACLF who are still graded as 2 or 3 after active medical treatment and/or artificial liver therapy, and the CLIF-C score is less than 64 points, it is recommended to perform liver transplantation as soon as possible within 28 days. Early liver transplantation is crucial for improving the prognosis of ACLF, reducing the risk of postoperative infection, progression from early ACLF to late ACLF, and further improving the 1-year post-transplant survival. The current priority for liver allocation based on MELD-Na can't give priority to liver donor matching to ACLF 1-2. Therefore, expanding the donor liver pool is an urgent need for early treatment of patients with ACLF. France team reviewed the development of APOLT to RAPID technology in liver transplantation for liver cirrhosis. Among them, 9 cases underwent two-step hepatectomy (including 5 cases of orthotopic assisted liver transplantation and 4 cases of RAPID surgery), 8 patients survived until the end of follow-up. Based on the experience of clinical practice, our center proposes and designs a clinical study of sequential adult left lateral lobe liver transplantation (SALT) for the treatment of early ACLF (Grade 1 and 2). On the basis of APOLT and RAPID, the safety and efficacy of sequential adult left lateral lobe liver transplantation were evaluated for the above patients.

DETAILED DESCRIPTION:
Acute on chronic liver failure (ACLF) is a type of liver failure that was considered an independent disease in 1995. It causes acute liver injury on the basis of chronic liver disease, leading to accelerated progression of existing liver diseases and liver failure. A meta-analysis of 30 global cohort studies using the EASL-CLIF C ACLF diagnostic criteria. Among 184041 patients with decompensated liver cirrhosis, the estimated prevalence of ACLF was 35%, and the estimated 90-day mortality rate was 58%.

ACLF is a syndrome characterized by rapid deterioration of liver function in chronic liver disease or undiagnosed chronic liver disease, with a short-term high risk of death. A retrospective study of 71894 hospitalized patients in the United States found that among the decompensated patients with liver cirrhosis, 18979 (26.4%) patients met the diagnosis of ACLF, with a 90-day mortality rate of 40%. Among them, ACLF grade 1 was 30.8%, grade 2 was 41.6%, and grade 3 was 68.8%. The Liver Failure and Artificial Liver Group of the Infectious Disease Branch of the CMA and the guidelines of EASL both mentioned that there is currently lack of specific drugs and methods for treatment of liver failure, mainly early diagnosis and treatment, dynamic evaluation; For patients with ACLF who are still graded as 2-3 levels after active treatment and/or artificial liver support, if the CLIF-C score is less than 64 points, it is recommended to perform liver transplantation as soon as possible within 28 days. According to the research of the Chinese severe hepatitis B research group, in patients with hepatitis B related ACLF, the survival rate at 28 days after transplantation was 86.9%, and the non-transplantation survival rate after matching analysis was 42.7%; The 90-day survival rate after transplantation is 82.5%, and the non-transplant survival rate is 32.1%; The one-year survival rate after transplantation is 77.2%, and the non-transplant survival rate is 27.6%. Therefore, liver transplantation is currently the only effective and definitive treatment for ACLF.

The mortality rate of 18416 ACLF patients waiting for liver transplantation in UNOS database is 21.6%. The waiting list mortality rates for ACLF grade 1, 2, 3a, and 3b are 18%, 20%, 25%, and 39%, respectively. The dynamic changes in ACLF patients during the waiting process for transplantation significantly affect their prognosis. The 1-year survival rate of ACLF transplant recipients who worsened from grade 0-2 to grade 3 was 83.8%, significantly lower than that of patients still in grade 0-2 (90.2%); When patients improve from grade 3 to grade 0-2 through medical treatment, the risk of mortality within 1 year after transplantation is reduced by 35%; Improved shock or severe hepatic encephalopathy, and ventilator removal are independent risk factors for decreased mortality after transplantation. In addition, the main factors for death within 1 year after ACLF transplantation are infection, and the 1-year survival rate of grade 3 ACLF patients significantly decreased (67.7%) after transplantation, while there was no significant difference in 5-year survival rate after 1 year. Wang et al reported that living donor liver transplantation has also achieved good results in the treatment of chronic and acute liver failure, with an average GRWR of 0.99 and a 3-year survival rate of 95.5%. Therefore, early liver transplantation is crucial for improving the prognosis of ACLF, reducing the risk of postoperative infection and progression from early ACLF to late ACLF, and further improving the 1-year survival rate.

As a reference score for organ allocation systems, only 9.1% of ACLF patients have a median MELD-Na score of 35. Therefore, ACLF patients should be transferred to transplant centers for evaluation as soon as possible; Further analysis revealed that in the MELD Na ≤9 group, the 90-day predicted mortality rate was 1.9%, while the actual mortality rates in ACLF grade 1 and 2 were 27.1% and 47.8%; In the MELD-Na 10-19 group, the 90-day predicted mortality rate was 6%, and the ACLF grade 1 and 2 mortality rates were 28.1% and 44.9%; In the MELD-Na group with a score of 20 or more, the 90-day predicted mortality rate is similar to the actual mortality rate, so the MELD-Na≤ 19 group severely underestimated the 90 day mortality rate of ACLF. Patients with ACLF grade 3 are highly susceptible to death or loss of transplant opportunities due to worsening conditions, especially those with MELD-Na scores lower than 25 in ACLF grade 3 patients, who do not have priority access to liver donors under the current allocation system. Therefore, the current priority scheme for liver allocation based on MELD-Na cannot give priority to liver source matching opportunities to ACLF grade 1-2 patients.

Therefore, expanding the donor liver pool is an urgent need for early treatment of patients with chronic and acute liver failure. Under normal circumstances, the graft receptor mass ratio (GRWR) needs to be greater than 0.8% in living donor liver transplantation or split liver transplantation, so adults often need half liver or more, increasing the risk of living donor and limiting the source of donors. In 2015, Line proposed a new surgical approach, which involves resection and partial liver segment (2-3 segments) transplantation combined with delayed total hepatectomy (RAPID) . This method can effectively avoid the waste of some livers without suitable child receptors. Therefore, it is possible to intentionally transplant the left lateral lobe (2+3 segments) to an adult recipient, while the remaining expanded right half liver is transplanted to another adult recipient. Compared to receiving whole liver transplantation, recipients receiving expanded right half liver transplantation did not suffer significant damage. Therefore, if RAPID surgery is confirmed to be feasible, it can greatly alleviate the problem of liver shortage in unresectable liver cancer, iCRLM, and ESLD patients, and improve the overall prognosis of these patients. The selection of liver donor sources can also consider adult live donor in addition to cadaver sources, as smaller 2+3 segments also have a smaller burden on the donor. In 2021, Balci group of Ankara University successfully treated a patient with liver cirrhosis, liver cancer and portal hypertension by using live RAPID. The GRWR was 0.42%. Two step surgery was performed in 35 days, and the patient was recovered and discharged 2 weeks later. Recently, Professor Scatton's team from France reviewed the development of APOLT to RAPID technology in liver transplantation for liver cirrhosis. Among them, 9 cases underwent two-step hepatectomy (including 5 cases of orthotopic assisted liver transplantation and 4 cases of RAPID surgery), with an 18-90 day interval between the first and second steps. The graft recipient body weight ratio ranged from 33% to 156%, and 1 patient died due to pulmonary infection after the second step surgery, One patient was unable to undergo two-step surgery due to biliary complications, and ultimately underwent whole liver orthotopic liver transplantation. All other 8 patients survived until the end of follow-up.

In summary, based on clinical surgical experience, our center proposes and designs a clinical study on Sequential Adult Left Lateral Segment Liver Transplantation (SALT), which involves assisted liver transplantation, portal inflow modulation, and two-stage hepatectomy for the treatment of early chronic acute liver failure. On the basis of APOLT and RAPID, the effectiveness and incidence of complications of were evaluated by sequential adult left lateral lobe liver transplantation (SALT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Diagnosed as acute-on-choronic liver failure according to APASL definition
* The severity of chronic and acute liver failure is diagnosed as level 1-2 according to the CANONIC criteria
* Signed informed consent and expected cooperation of the patients for treatment and follow up.

Exclusion Criteria:

* Clinical Frailty Scale score ≥ 7 points
* Severe hepatopulmonary syndrome, moderate to severe portal pulmonary hypertension; Surgical procedures with high risk of cardiovascular and pulmonary diseases
* Complicated with sepsis, various site infections such as spontaneous peritonitis, biliary tract infections, lung infections, bloodstream infections, urinary system infections, etc., did not improve after 72 hours of anti infection before transplantation; Gram negative bacterial infections resistant to carbapenems within the past 3 months
* Grade III-IV hepatic encephalopathy (West Haven classification), shock (with a dose of more than 1ug/Kg/min for demethylated kidney), PaO2/FiO2 value ≤ 150mmHg, renal failure requiring dialysis treatment
* Lactic acid greater than 9umol/L
* Special types of anatomical variations (such as portal vein III-IV type, etc.)
* Severe mental and psychological disorders
* Complicated with other diseases such as AIDS or malignant tumors
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 1 year after second stage hepatectomy
  To describe overall survival in patients with ACLF treated with sequential adult left lateral lobe liver transplantation.

SECONDARY OUTCOMES:
Graft Survival (GS) | 1 year after second stage hepatectomy
  To describe graft survival in patients with ACLF treated with sequential adult left lateral lobe liver transplantation
Postoperative complications | 90 days after liver transplant
  Describe the postoperative complications of sequential adult left lateral lobe liver transplantatiyn surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zhang, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No